CLINICAL TRIAL: NCT01236963
Title: Comparison of Efficacy on Interproximal Gingivitis and Dental Plaque Accumulation of an Essential Oils Mouthrinse and Dental Floss.
Brief Title: Essential Oils Mouth Rinse and Dental Floss: Efficacy on Interproximal Gingivitis and Dental Plaque Accumulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lisbon (Other)
Collaborators: Instituto Piaget (Other)
Responsible Party: Principal Investigator, Henrique Soares Luis, Professor, University of Lisbon
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 9/2006b
Record Dates: First submitted 2010-11-08; First posted 2010-11-09 (Estimated); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Gingivitis; Dental Plaque Accumulation
Keywords: Clinical trial; Prevention mouthrinse; Dental Floss
MeSH Terms: conditions — Gingivitis | interventions — Dental Devices, Home Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Essential oils mouthrinse (Experimental): Subjects use the essential oils mouthrinse
  Interventions: Drug: Essential oils mouthrinse
- Dental floss (Active Comparator): Subjects use dental floss
  Interventions: Device: Dental Floss

INTERVENTIONS:
Drug: Essential oils mouthrinse — Commercial mouthrinse with manufacturer's use indications
  Other Names: Listerine Cool Mint
  Arms: Essential oils mouthrinse
Device: Dental Floss
  Other Names: Colgate Total dental floss
  Arms: Dental floss

SUMMARY:
It is difficult to obtain patient's compliance with regular interproximal dental hygiene. Dental floss is recognized as an effective procedure to remove dental plaque and prevent gingivitis in the space between teeth, but it is difficult to use and most patients do no do it regularly. Essential oils mouthrinse acts on dental plaque bacteria and helps on gingivitis prevention. These properties may be of interest to control dental plaque accumulation and gingivitis in interproximal areas. The study hypothesis states that there are no differences between the use of an essential oils mouthrinse and dental floss on the reduction of dental plaque accumulation and gingivitis.

DETAILED DESCRIPTION:
The use of mouthwashes or rinses as an adjunct to mechanical plaque removal should be considered by oral health professionals as part of a strategy to prevent and control patients' oral problems. Most individuals do not brush or floss for the required duration or with the necessary skill to ensure effectiveness, even after receiving hygiene instruction and motivation (Beals et al., 2000; Ciancio, 2003; Santos, 2003). Consequently, inadequate oral hygiene leads to plaque buildup, a key etiological factor in periodontal disease and dental caries. Mouthwashes containing essential oils and rinses with delmopinol have proven effective in controlling plaque development and preventing gingivitis (Baehni and Takeuchi, 2003).

The American Dental Association (ADA) has established guidelines for studying the efficacy of oral hygiene products on gingivitis and plaque accumulation. These guidelines, found in the Acceptance Program Guidelines, provide instructions on planning and evaluating various types of laboratory and clinical studies to test mouthwashes and rinses (ADA, 1997-2008).

In laboratory studies, the effectiveness of antiseptic oral products is tested for their ability to inhibit oral microorganisms. The goal is to determine if these products alter the oral flora. Plaque samples for these studies are collected at baseline and at the end of the experimental period from a predetermined dental surface. Samples are recorded in colony-forming units per millilitre (CFU/ml). For non-specific plaque evaluation, samples are grown on a general nutrient medium, while specific bacteria require selective culture media (ADA, 2008). Bacterial resistance and growth inhibition are assessed using the minimum inhibitory concentration method, typically via the disk diffusion test (ADA, 2008).

Clinical studies, approved by an ethics committee, must demonstrate the efficacy of mouthwashes and rinses in reducing plaque accumulation and gingivitis. Participants undergo a comprehensive oral examination at the study's outset to assess initial conditions, inclusion, and exclusion criteria, and to obtain informed consent (ADA, 1997). Clinical variables are measured at baseline, at study end, and optionally at an intermediate point (ADA, 2006). Sample size must allow for statistical testing with a significance level of 1% or 5% and a power of 80% whenever possible (ADA, 2007). Study duration varies by objective; demonstrating antiseptic properties requires at least six months, while evaluating effects on gingivitis and plaque can be done in as little as two weeks (Collaert et al., 1992-2007).

Participants should be from the product's target population, with usage not necessarily supervised by the researcher. Studies must include both genders and various age groups, with random assignment to experimental and control groups (ADA, 2008). Participants must be healthy adults with no oral pathology and similar oral hygiene conditions, avoiding medications that affect gingival parameters during the study (ADA, 2008). Clinical variables related to plaque and gingivitis are assessed using scientifically recognized indices.

In summary, this study aims to evaluate the effectiveness of mouthwashes and rinses in controlling plaque and gingivitis, following established guidelines to ensure rigorous and systematic assessment.

ELIGIBILITY:
Inclusion Criteria:

* To be a student at the Dental Hygiene programme at the Lisbon Dental School
* Signature on informed consent form
* Have, at least, two quadrant with 6 teeth each
* Presence of dental plaque

Exclusion Criteria:

* Use of a mouthrinse
* Dental hygiene appointment in the past 6 months
* Use of antibiotics in the past 3 months
* Presence of extensive caries and fractures of teeth

Ages: 15 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2007-09; Primary Completion 2008-01 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Lobene Gingival Index | change from baseline in gingival index at two weeks
  data collected at the begining of the study and two weeks after mouthrinse or dental floss use
Saxton & Ouderaa Bleeding Index | change from baseline in bleeding index at two weeks
  data collected at the begining of the study and two weeks after mouthrinse or dental floss use
Quigley, Hein & Turesky Dental Plaque Index | change from baseline in plaque index at two weeks
  data collected at the begining of the study and two weeks after mouthrinse or dental floss use

CONTACTS AND LOCATIONS:
Overall Officials: Mario F Bernardo, PhD, Study Director — Faculdade de Medicina Dentária da Universidade de Lisboa
Locations (1):
- Faculdade de Medicina Dentária da Universidade de Lisboa, Lisbon, Portugal

REFERENCES:
- [Background] Barnett ML. The rationale for the daily use of an antimicrobial mouthrinse. J Am Dent Assoc. 2006 Nov;137 Suppl:16S-21S. doi: 10.14219/jada.archive.2006.0408. PMID 17035671
- [Background] Bauroth K, Charles CH, Mankodi SM, Simmons K, Zhao Q, Kumar LD. The efficacy of an essential oil antiseptic mouthrinse vs. dental floss in controlling interproximal gingivitis: a comparative study. J Am Dent Assoc. 2003 Mar;134(3):359-65. doi: 10.14219/jada.archive.2003.0167. PMID 12699051
- [Background] Gordon JM, Lamster IB, Seiger MC. Efficacy of Listerine antiseptic in inhibiting the development of plaque and gingivitis. J Clin Periodontol. 1985 Sep;12(8):697-704. doi: 10.1111/j.1600-051x.1985.tb00941.x. PMID 3902908
- [Background] Sharma N, Charles CH, Lynch MC, Qaqish J, McGuire JA, Galustians JG, Kumar LD. Adjunctive benefit of an essential oil-containing mouthrinse in reducing plaque and gingivitis in patients who brush and floss regularly: a six-month study. J Am Dent Assoc. 2004 Apr;135(4):496-504. doi: 10.14219/jada.archive.2004.0217. PMID 15127875
- [Background] Sharma NC, Charles CH, Qaqish JG, Galustians HJ, Zhao Q, Kumar LD. Comparative effectiveness of an essential oil mouthrinse and dental floss in controlling interproximal gingivitis and plaque. Am J Dent. 2002 Dec;15(6):351-5. PMID 12691269